CLINICAL TRIAL: NCT00415753
Title: Procalcitonin as a Marker of Bacterial Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Skejby Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 271-05-0765
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Pneumonia; Bronchitis; COPD
MeSH Terms: conditions — Pneumonia; Bronchitis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: No antibiotics if se-procalcitonin is below stated limit

SUMMARY:
Objective: To evaluate PCT as a marker of bacterial community acquired pneumonia in a Danish Hospital setting. To test if it is possible to reduce the use of antibiotics and the length of stay in hospital, and the willingness of the clinicians to take this new marker under advisement in their choice of treatment.

The study is a randomised, controlled intervention study. All adult patients admitted to the Department of Infectious Disease at Skejby hospital suspected of a lower respiratory tract infection (e.g. CAP, acute exacerbation of COPD and bronchitis) are eligible for inclusion. Patients are randomised to have either PCT guided treatment or standard care, in which case the doctor will not learn the PCT test result. In the PCT group the antibiotic treatment will be based on serum PCT as follows: If PCT is less than 0.25 µg/L antibiotic treatment is discouraged; if PCT is greater than 0.25 µg/L antibiotic treatment is encouraged and if PCT is greater than 0.5 µg/L antibiotic treatment is strongly encouraged. The treating doctor is allowed to overrule the treatment guidelines. The control group will receive antibiotics according to usual practice.

The primary endpoints are antibiotic use and length of stay in hospital. Secondary endpoint is the proportion of patients where the treating doctor chooses to disregard the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* suspected lower respiratory tract infection
* must be able to give consent

Exclusion Criteria:

* age under 18 years
* not able to give consent
* admitted not primarily because of the respiratory tract infection
* hospital acquired infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Antibiotic use
Length of stay in hospital

SECONDARY OUTCOMES:
The proportion of patients where the doctor chooses to disregard treatment guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Finn T Black, Professor, Study Chair — Aarhus Universityhospital; Kristina B Kristoffersen, Principal Investigator — Aarhus University Hospital Skejby
Locations (2):
- Denmark (2):
  - Department of Infectious Diseases, Skejby Hospital, Aarhus N
  - Departement of Medicin, Silkeborg Hospital, Silkeborg

REFERENCES:
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Derived] Kristoffersen KB, Sogaard OS, Wejse C, Black FT, Greve T, Tarp B, Storgaard M, Sodemann M. Antibiotic treatment interruption of suspected lower respiratory tract infections based on a single procalcitonin measurement at hospital admission--a randomized trial. Clin Microbiol Infect. 2009 May;15(5):481-7. doi: 10.1111/j.1469-0691.2009.02709.x. Epub 2009 Mar 5. PMID 19416298